CLINICAL TRIAL: NCT04837742
Title: The Effect of Ultrasound-guided Erector Spinae Plane Block on Postoperative Analgesia in Radiofrequency Ablation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202101007RINA
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; radiofrequency ablation; erector spinae plane block
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Experimental): ESPB injection at T10 region with levobupivacaine 100mg (20 ml)+ Omnipaque10 ml
  Interventions: Drug: ESPB group
- Control group (Sham Comparator): ESPB injection at T10 region with 0.9% normal saline 20ml + Omnipaque10ml
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: ESPB group — ESPB injection at T10 region with Chirocaine 100mg(20 cc)+ Omnipaque 10cc
  Arms: ESPB group
Drug: Control group — ESPB injection at T10 region with Normal saline 20cc + Omnipaque 10cc
  Other Names: ESPB group
  Arms: Control group

SUMMARY:
This is a double blind, randomized controlled trial to evaluate the efficacy of ESPB(Erector Spinae Plane Block) on postoperative analgesia in RFA( Radiofrequency Ablation therapy). We will include 80 patients, and randomly assign to ESPB(Chirocaine) group and control group(normal saline).We deduce Erector spinae plane block can be use as a postoperative analgesic way for patients who receive radiofrequency ablation of hepatocellular carcinoma.

DETAILED DESCRIPTION:
Computed tomography guided radiofrequency ablation of hepatocellular carcinoma(HCC) has became a popular way to treat HCC. Although the wound is small and the patients can discharge on the next day, they have to suffer from moderate to severe pain. Nowadays Erector spinae plane block has been applied to many surgery as a postoperative analgesic strategy. We deduce Erector spinae plane block can be use as a postoperative analgesic way for patients who receive radiofrequency ablation of hepatocellular carcinoma. Besides, we will add contrast medium to evaluate the spread area of local anesthetics.

ELIGIBILITY:
Patients undergoing computed tomography guided radiofrequency ablation of hepatic tumor under scheduled general anesthesia, and fulfilled one of following inclusion criteria:

1. diameter of hepatic tumor is larger than 2 cm
2. distance of tumor site is near the hepatic surface < 2cm

Exclusion criteria:

1. A history of allergic reaction to local anesthetics or iohexol
2. Renal insufficiency, creatinine clearance < 30mL/min
3. Coagulopathy or other bleeding disorder that cannot perform nerve block
4. Under pregnancy or lactation
5. Opioid tolerant patient

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scale at postoperative day one | approximately 12-24 hrs
  We will assess the pain intensity by using a 100-mm visual analogue scale at postoperative day one
Drug spread level of erector spinae plane block | approximately 2-3 hrs
  We will assess the numbers of vertebral levels of erector spinae block drug spreading by using computed tomography

SECONDARY OUTCOMES:
Visual analogue pain scale at post-anesthesia care unit | approximately 3 hours
  We will assess the pain intensity by using a 100-mm visual analogue scale at post-anesthesia care unit
Postoperative recovery quality | approximately 2 days
  We will assess the quality of recovery by using QoR-15 questionnaire at the postoperative day one

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan